CLINICAL TRIAL: NCT01403480
Title: Rates of Positive BCCs in Re-excisions
Brief Title: Rates of Positive Basal Cell Carcinomas (BCCs) in Re-excisions
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Yehuda Ullmann, Head, Plastic and Reconstructive Surgery Department, Rambam Healthcare Campus
Other Study IDs: 0064-11-RMB-CTIL
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-02

CONDITIONS: Basal Cell Carcinoma
Keywords: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Basal Cell Carcinoma (BCC) is the most common malignant growth in the world. Treatment is primarily surgical with the goal of excising the growth in its entirety. When pathology results show that this has not been achieved, a re-excision is routinely performed. This study examines retrospectively the percentage of re-excisions of BCC that actually proved to be positive (exhibited growth) among those re-excisions performed at Rambam Healthcare Campus and Zvulun Community Medical Center during the years 2008-10.

ELIGIBILITY:
Inclusion Criteria:

All patients that underwent an incomplete BCC excision during the years 2008-2010.

Exclusion Criteria:

Patients that underwent an incomplete BCC excision and were subsequently referred to undergo a MOHS procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that underwent an incomplete BCC excision during the years 2008-2010.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)